CLINICAL TRIAL: NCT02419716
Title: A Longitudinal Study of Cologuard™ in an Average Risk Population Assessing a Three Year Test Interval
Brief Title: A Study of Cologuard™ in an Average Risk Population Assessing a Three Year Test Interval
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Exact Sciences 2014-01
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer Screening; Colorectal Cancer
Keywords: colorectal cancer; Colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A portion of the stool sample may be retained, if any remains after the study-related tests for use in a sample bank for use in the future. The samples may be stored for up to twenty (20) years. These stool samples will de-identified.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cologuard — Prescription of Cologuard for at-home stool collection

SUMMARY:
This is a prospective longitudinal study to assess the impact of repeat Cologuard testing at 3 years in average risk patients.

DETAILED DESCRIPTION:
This is a prospective longitudinal study to assess the impact of repeat Cologuard testing at 3 years in average risk patients. Enrolled subjects will be prescribed Cologuard per approved labeling at baseline. Subjects with positive results will be referred to colonoscopy and study participation completed. Subjects with negative Cologuard results will be seen annually for 3 years. At year 3, subjects will repeat Cologuard, followed by colonoscopy, regardless of the Cologuard test outcome. Subjects who have a colonoscopy at any time during the study will be discontinued following collection of the colonoscopy and associated histopathology results.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been prescribed Cologuard for colorectal cancer screening
2. Subject is at average risk for development of colorectal cancer
3. Subject is 50 years or older
4. Subject willing and able to sign informed consent.

Exclusion Criteria:

1. Subject had a colonoscopy in the previous 9 years
2. Subject has undergone any double-contrast barium enema, virtual (CT-based) colonoscopy, or flexible sigmoidoscopy within the previous five (5) years.
3. Subject has had a positive fecal occult blood test or FIT within the previous six (6) months.
4. Subject has any condition that in the opinion of the investigator should preclude participation in the study (e.g., subject not eligible for a diagnostic colonoscopy).
5. Subject has a history of colorectal cancer or advanced adenoma.
6. Subject has a history of aerodigestive tract cancer
7. Subject has had a prior colorectal resection for any reason other than sigmoid diverticular disease
8. Subject has had overt rectal bleeding, e.g. hematochezia or melena, within the previous 30 days. (Blood on toilet paper, after wiping, does not constitute rectal bleeding)
9. Subject has a diagnosis or personal history of any of the following high-risk conditions for colorectal cancer:

   * Inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease.
   * 2 first-degree relatives who have been diagnosed with colon cancer. (Note: first-degree relatives include parents, siblings and offspring).
   * One first-degree relative with CRC diagnosed before the age of 60.
10. Subject has a family history of:

    * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP).
    * Hereditary non-polyposis colorectal cancer syndrome (also referred to as "HNPCC" or "Lynch Syndrome").
    * Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Gardner's Syndrome, Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Cronkhite-Canada Syndrome, Neurofibromatosis and Familial Hyperplastic Polyposis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll approximately 2,400 men and women aged 50 years and older at a minimum of 20 sites to achieve a minimum of 1,119 subjects at the Year 3 visit. To increase the point prevalence of CRC in the study population, subject enrollment will be age-weighted toward a slightly older population. Enrollment of at least 65% of subjects age 65 years or older will be targeted
Sampling Method: Non-Probability Sample
Enrollment: 2404 (Actual)
Dates: Start 2015-04; Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Predictive Value | Three years
  The difference between the positive predictive value (PPV) at year 3 (PPV3) and 1 minus the negative predictive value (NPV) at year 3 (NPV3).

SECONDARY OUTCOMES:
Colorectal Cancer Incidence | 3 years
  Observed versus the expected reduction in colorectal cancer incidence at year 3 (T3)

OTHER OUTCOMES:
Predictive value of a positive Cologuard result at baseline (T0) | baseline
  Predictive value of a positive Cologuard result at baseline (T0)
The predicative value of a positive and a negative Cologuard at year 3 (T3). | 3 years
  The predicative value of a positive and a negative Cologuard at year 3 (T3).
The sensitivity and specificity of Cologuard at year 3 (T3). | 3 years
  The sensitivity and specificity of Cologuard at year 3 (T3).
The positive (PLR) and negative (NLR) likelihood ratios at year 3 (T3). | 3 years
  The positive (PLR) and negative (NLR) likelihood ratios at year 3 (T3).
The cumulative risk of false positive result (cFPR) and cumulative risk of a true positive result (cTPR). | 3 years
  The cumulative risk of false positive result (cFPR) and cumulative risk of a true positive result (cTPR).
The probability that a negative Cologuard result at baseline remains negative through 3 years. | 3 years
  The probability that a negative Cologuard result at baseline remains negative through 3 years.
The probability that a negative Cologuard result at baseline (T0) results in no CRC/AA through 3 years. | 3 years
  The probability that a negative Cologuard result at baseline (T0) results in no CRC/AA through 3 years.
The distribution of colorectal epithelial lesions (by Category) among positive Cologuard subjects at T0 and at T3 | 3 years
  The distribution of colorectal epithelial lesions (by Category) among positive Cologuard subjects at T0 and at T3
Adherence to repeat Cologuard at year 3 (T3) | 3 years
  Adherence to repeat Cologuard at T3 will be reported with counts and proportions.
Compliance to colonoscopy following a positive Cologuard result | baseline
  Cumulative compliance to colonoscopy following a positive Cologuard result
Cross-over to alternative screening methodologies (e.g. FOBT, colonoscopy, other) at T1,T2, and T3 | Years 1, 2, and 3
  Cross-over to alternative screening methodologies (e.g. FOBT, colonoscopy, other) at T1,T2, and T3
The rate of no Cologuard result (e.g. invalid result) | 3 years
  The rate of no Cologuard result (e.g. invalid result)
The adverse event rate (events occurring between collection kit distribution and sample submission) | 3 years
  The adverse event rate (events occurring between collection kit distribution and sample submission)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Imperiale, MD, Principal Investigator — Indiana University
Locations (40):
- United States (40):
  - Thomas C Lenzmeier, M.D., P.C, Glendale, Arizona
  - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Cassidy Medical Group/Radiant Research, Inc., Carlsbad, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Paragon Rx Clinical, Garden Grove, California
  - UCLA, Division of Digestive Diseases, Los Angeles, California
  - FACEY Medical Foundation, Mission Hills, California
  - John D. Homan, MD, Newport Beach, California
  - Diverse Research Solutions, Oxnard, California
  - Ventura County Gastroenterology, Oxnard, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Advanced Pain Diagnostics & Solutions, Sacramento, California
  - Innovative Research of West Florida, Clearwater, Florida
  - Homestead Medical Research, Homestead, Florida
  - Health Awareness, Inc, Jupiter, Florida
  - Precision Clinical Research, Lauderdale Lakes, Florida
  - Advanced Bioresearch, Miami, Florida
  - Next Phase Research Alliance, Miami, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Health Awareness, Inc-Port St. Lucie, Port Saint Lucie, Florida
  - The Kaufmann Clinic, Inc., Atlanta, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Pharmakon Inc, Evergreen Park, Illinois
  - Indiana University, Eskanazi Hospital, Regenstrief Health Center, Indianapolis, Indiana
  - MedPharmics, LLC, Metairie, Louisiana
  - Columbia Medical Practice, Columbia, Maryland
  - Centennial Medical Associates, Elkridge, Maryland
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Nevada Family Care, Henderson, Nevada
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Sentral Clinical Research, Cincinnati, Ohio
  - Comprehensive Internal Medicine, Inc., Wooster, Ohio
  - Family Practice Center of Wooster, Inc./Clinical Trial Developers, Wooster, Ohio
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Austin Regional Clinic, Austin, Texas
  - PCP for Life (DM Research), Montgomery, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include text, tables, figures, and appendices. The study protocol, statistical analysis plan, informed consent form, and clinical study report will also be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from 2 years and ending 4 years after publication. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will be available between 2 and 4 years after publication through the Sponsor.